CLINICAL TRIAL: NCT03466684
Title: Bioelectrical Impedance Analysis Guided-Fluid Management Promotes Primary Fascial Closure of Postinjury Open Abdomen
Brief Title: BIA Guided-fluid Management in Postinjury Open Abdomen
Acronym: BGFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Clinical Professor, Nanjing PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012NLY096
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-03

CONDITIONS: Damage Control; Trauma Abdomen; Acute Compartment Syndrome
Keywords: Trauma; Open abdomen; Fluid resuscitation; Fascial closure; Bioelectrical impedance analysis
MeSH Terms: conditions — Abdominal Injuries; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIA-directed fluid resuscitation (Experimental): After the achievement of CVP, MAP and ScvO2 goals, if hyperhydration (HL > 74.3%) was found, then the following fluid management was applied with each passing 6h. If HL was above 87% (severe level), fluid infusion was restricted, a furosemide drip was used, and CRRT was initiated with an ultrafiltration rate when patients were failure or inadequate response to above diuretic therapy that gave a net negative fluid balance of at least 1500 ml during the next 6h. If HL was 81%-87% (moderate level), above methods were used to trigger a net negative fluid balance (about 1000 ml) for the next 6h. Similarly, If HL was 74.3%-81% (mild level), a net negative fluid balance of about 500 ml would be achieved during the next 6h of ICU hospitalization. If HL was blow 71%, a state of dehydration, CVP, MAP, and ScvO2 was maintained as above during ICU resuscitation.
  Interventions: Other: BIA-guided fluid resuscitation protocol
- Traditional fluid resuscitation (Active Comparator): A timely restricted intravenous fluid regimen or dehydration therapy was implemented by two senior clinicians according to cumulative fluid balance recording and hemodynamic condition such as heart rate, blood pressure, central venous pressure, mean arterial pressure, urine output and body weight change.
  Interventions: Other: Traditional fluid resuscitation protocol

INTERVENTIONS:
Other: BIA-guided fluid resuscitation protocol — In both groups, a multi-frequency BIA with eight tactile electrodes (Inbody S10 Biospace, Biospace Co. Ltd., Seoul, Korea) was used to assess body fluid status every 6h within the first 72h after admission to the ICU and daily for a period of 4 days.
  BIA recording was not adjusted by clinicians in fluid restrict, pharmacological and mechanical means of therapy.
  In contrast, in group BIA, fluid resuscitation protocol with adjustment determined according to HL measured by BIA.
  Arms: BIA-directed fluid resuscitation
Other: Traditional fluid resuscitation protocol — Traditional fluid resuscitation strategy determined by treating clinicians according to usual clinical parameters.
  Arms: Traditional fluid resuscitation

SUMMARY:
Fluid overload (FO), resulting from high volume fluid therapy, is frequent and contributes to excessive visceral edema, delayed fascial closure, and adverse outcomes among postinjury open abdomen (OA) patients. Bioelectrical impedance analysis (BIA) is a promising tool in monitoring fluid status and FO. Thus, we sought to investigate the efficacy of BIA-directed resuscitation among postinjury OA patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients admitted to SICU with OA after emergent abbreviated laparotomy were considered eligible.

Exclusion Criteria:

* (a) age less than 18 years; (b) pregnancy; (c) lactation; (d) limb amputations; (e) mental disorders; (f) diabetes mellitus; (g) pre-existing blood disorders; (h) pre-existing abdominal fistulas; (i) pre-existing terminal illness; (j) liver dysfunction (Child-Pugh class C); (k) New York Heart Association (NYHA) class IV; (l) chronic renal failure requiring dialysis; (m) therapy with an extra-corporeal membrane oxygenator (ECMO); (n) enrolled in an ongoing, interventional RCT; (o) received prior fluids for resuscitation during their ICU stay; (p) expected to die within 1 hour of ICU admission for devastating injuries; (q) activated opt-out process for BGFM trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of 30-day primary fascial closure | 30 days
  Rate of 100% direct approximation of abdominal fascial edges

SECONDARY OUTCOMES:
Time to fascial closure | 30 days
  Time to 100% direct approximation of abdominal fascial edges
Postoperative 7-day fluid volume | 7 days
  Statistics of postoperative 7-day fluid volume Postoperative 7-day fluid fluid use during resuscitation
Postoperative 30-day mortality | 30 days
  All cause mortality within 30 days
Postoperative 30-day adverse effects | 30 days
  All cause adverse effects within 30 days